CLINICAL TRIAL: NCT05489523
Title: An Open-label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Tafamidis in Patients With Transthyretin-mediated Amyloidosis Post Orthotopic Heart Transplantation
Brief Title: Safety, Efficacy, and Pharmacokinetics of Tafamidis in Patients With Transthyretin-mediated Amyloidosis Post Orthotopic Heart Transplantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Justin Grodin, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0583
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Transthyretin Cardiac Amyloidosis
Keywords: heart transplantation; transthyretin amyloidosis; ATTR; tafamidis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Tafamidis 61 mg
  Interventions: Drug: Tafamidis 61 MG

INTERVENTIONS:
Drug: Tafamidis 61 MG — Tafamidis 61 mg by mouth daily for 12 months

SUMMARY:
Transthyretin cardiac amyloidosis (ATTR-CA) is a relentlessly progressive disease that can progress to end stage heart failure, at which point recently approved transthyretin production silencing or structure stabilizing therapies provide no clinical benefit. For well-selected individuals, heart transplantation is an excellent therapeutic option to improve survival. Historically, concomitant liver transplantation has been used to halt the progression of non-cardiac transthyretin amyloidosis (ATTR) manifestations, especially for individuals with TTR genotypes associated with significant neuropathy. However, despite this, patients continue to experience progressive non-cardiac manifestations, particularly gastrointestinal and neuropathic, which can have a substantial influence on post-heart transplantation morbidity. Concomitant liver transplantation is also associated with substantial morbidity and its future therapeutic role is questionable with recently established therapies for ATTR. Therefore, there is a clear unmet need to determine the utility and safety of ATTR targeted therapies for patients with recent heart transplantation for end-stage ATTR-CA. The central hypothesis of this proposal is that in patients who have received a heart transplantation for end-stage ATTR-CA, tafamidis therapy will be efficacious and well-tolerated. We aim to determine the safety and efficacy of tafamidis in stable patients who have undergone heart or combined heart/liver transplantation for ATTR (wild-type or variant) cardiac amyloidosis. The proposed study will be a single-arm intervention clinical trial with tafamidis. Because of the efficacy of tafamidis for both variant ATTR-CA and wild-type ATTR-CA, there is no clinical equipoise for an inactive-comparator placebo arm. The primary endpoint of this study will be serial change in plasma transthyretin (TTR) levels from baseline to 12 months at 3-month intervals. The secondary endpoints of this study will include serial changes in neuropathy assessments, modified body mass indices, incident transplant-specific adverse events, and pharmacokinetics of tafamidis. Observations from this study will establish the role of tafamidis use for the management of ATTR in patients after transplantation for end-stage ATTR-CA.

DETAILED DESCRIPTION:
A. Primary Aim

To determine the safety and efficacy of tafamidis in patients who have undergone heart or combined heart/liver transplantation for ATTR (wild-type or variant) cardiac amyloidosis.

Primary Hypothesis. Initiation of the TTR stabilizer, tafamidis, post heart or heart/liver transplant for ATTR cardiac amyloidosis, (wild-type or variant disease) will be associated with an increase in plasma transthyretin levels during 12 months of therapy.

B. Secondary Aims

1. To determine the impact of tafamidis on serial questionnaire assessments that quantitate and determine the severity and clinical implications of motor, sensory, and autonomic neurologic impairment in participants over 12 months with cardiac transplantation.
2. To determine the impact of tafamidis on serial questionnaire assessment of activity and social participation limitation, dysautonomia and nutritional status in participants over 12 months with cardiac transplantation.
3. To determine the impact of tafamidis on transplantation-related adverse events in participants over 12 months with cardiac transplantation.
4. To establish the pharmacokinetics of tafamidis in participants with cardiac transplantation over 12 months.

C. Study Type / Design

The proposed study will be a single-arm, intervention clinical trial. Because of the observed efficacy of tafamidis and other therapies for both ATTRv and ATTRwt, there is no clinical equipoise for an inactive-comparator placebo arm.

D. Expected Outcomes

Upon completion of this clinical trial, it is our expectation that we will establish the efficacy and safety of tafamidis in patients with who have undergone heart transplantation for ATTR-CA. Further, we expect to have shown that tafamidis will have predictable pharmacokinetics and will lead to improvement in polyneuropathy questionnaire scores and mBMI. Such findings would be important, because they would justify the use of tafamidis to halt ATTR progression in patients who have undergone heart transplantation for advanced ATTR-CA.

Specifically, we will expect the following:

1. Tafamidis will be safe and well tolerated in the post heart transplant population, providing data to support its use as a therapeutic agent to halt the progression of extra cardiac manifestations of TTR amyloidosis post HT for end stage ATTR-CA.
2. TTR levels will increase from baseline at the 3-month visit and remain stable throughout the remainder of the study period. This increase in serum TTR will be comparable to that seen in the ATTR-ACT trial, reflective of stabilization of TTR and treatment efficacy in this patient population.
3. Serial assessment of Norfolk-QoL-DN, COMPASS-31 and R-ODS questionnaires will demonstrate stable disease at 12 months as measured by autonomic symptoms and quality of life.
4. There will be no increase, from baseline, in incidence of treated acute cellular rejection, antibody mediated rejection, active CMV infection, coronary allograft vasculopathy or post-transplant lymphoproliferative disorder as a result of concurrent TTR stabilizing therapy with tafamidis.
5. Plasma pharmacokinetics of tafamidis free acid in the post HT population will be similar to those observed in previous studies of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Has received orthotopic heart transplantation for end-stage ATTRv or ATTRwt ≥12 months prior to screening. Concomitant hepatic and renal transplantation with adequate allograft function are included.
* Has a stable immunosuppressive regimen and ≤ 10 mg of prednisone (or equivalent) at time of enrollment.
* Has a Karnofsky performance status ≥ 70%

Exclusion Criteria:

* Has previously received inotersen within the past 180 days, patisiran within the past 90 days, tafamidis within the past 14 days, or diflunisal in the past 14 days.
* Participating in a clinical trial for ATTR targeted therapies.
* Has an estimated glomerular filtration rate (eGFR) ≤ 15 ml/min/1.73 m2
* Has known leptomeningeal or AL amyloidosis
* Has active post-transplant lymphoproliferative disease
* Excluding non-melanomatous skin cancers, has an active malignancy.
* Has active infection with hepatitis B, hepatitis C, human immunodeficiency virus, or cytomegalovirus (CMV). For CMV, donor/ recipient exposure status and prior treated CMV disease on stable doses of antiviral therapies are not excluded.
* Has cardiac allograft dysfunction defined by left ventricular ejection fraction (LVEF) <50% by echocardiogram within the past 3 months
* Has been treated for acute cellular or antibody mediated rejection in the past 3 months
* Has criteria to meet International Society for Heart and Lung Transplantation standardized nomenclature for severe coronary allograft vasculopathy ("ISHLT CAV3")

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Serial change from baseline in plasma TTR levels at 12 months | Baseline, 3, 6, 9, and 12 months
  Serial change from baseline in plasma Time in Therapeutic Range (TTR) levels at 12 months is measured at 3 month intervals. TTR tetramer stability is measured using an immunoturbidimetric assay. Increase in plasma TTR levels indicate TTR tetramer stability.

SECONDARY OUTCOMES:
Serial change from baseline in Norfolk QoL-DN at 12 months | Baseline, 3, 6, 9, and 12 months
  Serial change from baseline in Norfolk Quality of Life Diabetic Neuropathy (QoL-DN) at 12 months is measured at 3 month intervals. The Norfolk-QoL-DN total score differentiates between healthy subjects and individuals with ATTRv polyneuropathy as well as different stages of Transthyretin amyloidosis (ATTR) polyneuropathy. The total score has a range of -4 to 136, with a higher score indicating worse disease symptoms. There are five different domains assessed within an overall quality of life score: symptoms, large fiber, small fiber, activities of daily living and autonomic dysfunction.
Serial change from baseline in Composite Autonomic Symptom Score (COMPASS-31) at12 months | Baseline, 3, 6, 9, and 12 months
  Serial change from baseline in Composite Autonomic Symptom Score (COMPASS-31) at12 months is measured at 3 month intervals. COMPASS-31 is a 31-question participant-reported assessment that measures autonomic symptoms across 6 weighted domains on a 100-point scale: orthostatic intolerance (40 points), vasomotor (5 points), secretomotor (15 points), gastrointestinal (25 points), bladder (10 points), and pupillomotor (15 points). A higher score indicates worse autonomic dysfunction.
Number of transplant-specific adverse events | 12 months
  Transplant-specific Adverse events will be determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Number of hepatic or renal transplant-specific adverse events | 12 months
  Hepatic or renal transplant-specific adverse events will be determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Steady-state plasma concentration of tafamidis in patients undergone HT for end stage ATTR-CA | Baseline, 3, 6, 9, and 12 months
  Steady-state plasma pharmacokinetic (PK) parameters will calculated based on plasma concentration of tafamidis in patients who have undergone HT for end stage ATTR-CA.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Grodin, MD, Principal Investigator — University of Texas Southwestern Medical Center; Jan Griffin, MD, Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - Cedars-Sinai, Beverly Hills, California
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No